CLINICAL TRIAL: NCT04479566
Title: Effect of Lithium Carbonate on Postoperative Sleep in Patients Undergoing Videoassisted Thoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-27-2
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2020-11

CONDITIONS: Sleep Deprivation
Keywords: bispectral index; lithium carbonate
MeSH Terms: conditions — Sleep Deprivation | interventions — Lithium Carbonate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lithium carbonate (Experimental): Patients undergoing video assisted thoracic surgery during the morning will take 250mg lithium carbonate 6 hours after surgery.
  Interventions: Drug: Lithium Carbonate 250 MG
- calcium carbonate (Placebo Comparator): Patients undergoing video assisted thoracic surgery during the morning will take calcium carbonate 500mg 6 hours after surgery.
  Interventions: Drug: Calcium Carbonate 500 MG

INTERVENTIONS:
Drug: Lithium Carbonate 250 MG — Patients undergoing video assisted thoracic surgery during the morning will take 250mg lithium carbonate 6 hours after surgery.
  Arms: lithium carbonate
Drug: Calcium Carbonate 500 MG — Patients undergoing video assisted thoracic surgery during the morning will take calcium carbonate 500mg 6 hours after surgery.
  Arms: calcium carbonate

SUMMARY:
It has been proved that lithium carbonate can prolong slow wave sleep with few or no side-effects. The aim of the present study is to evaluate postoperative sleep quality of patients undergoing video assisted thoracic surgery taken 250mg lithium carbonate 6 hours after surgery.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled (randomized, parallel group, concealed allocation), double-blinded trial. All patients undergoing video assisted thoracic surgery during morning will be randomized 1:1 to the treatment intervention with lithium carbonate 250mg (Baoqing, Hunan, China) or calcium carbonate 500mg (Reneed, Beijing, China) 6 hours after surgery. The objective of the trial is to evaluate the lithium carbonate 250mg on the first postoperative night sleep quality. The patients received standardized general anesthesia supplemented by paravertebral nerve block. The ultrasound-guided approach for paravertebral nerve block was used with the patient in the lateral decubitus position, and the paravertebral nerve block was administered at the T4-T6 level according to the incision protocol at our center. General anesthesia for maintenance of propofol anesthesia, total intravenous anesthesia was administered by using propofol (Fresenius Kabi, Austria GmbH) at a plasma target concentration (Marsh pharmacokinetic model software) of 2.5-4 μg/ml. Remifentanil (0.2-0.5 μg/kg/min, Renfu, Yichang, China) was given to all patients during the operation. All patients accepted patient-controlled intravenous analgesia with 1 μg ml-1 sufentanil (Renfu, Yichang, China). Duration of sleep was defined as the duration of all bispectral index data below 80 in the 12 hours of monitoring (from 20:00pm to 06:00am).

ELIGIBILITY:
Inclusion Criteria:

* • 1. ethnic Chinese;
* • 2. age, 18 to 75 years old;
* • 3. American Society of Anaesthesiologists (ASA) physical status I or II;
* • 4. required VATS for lung surgery and one lung ventilation

Exclusion Criteria:

* Cognitive difficulties
* • Partial or complete gastrectomy
* • Previous esophageal surgery
* • Previous treated by radiotherapy or surgery
* • Inability to conform to the study's requirements
* • body mass index exceeding 30 kg/m2
* • Deprivation of a right to decide by an administrative or juridical entity
* • Ongoing participation or participation in another study <1 month ago
* • preoperative Pittsburgh Sleep Quality Index global scores higher than 6
* • recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or traditional Chinese medicine

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 51 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
sleep quality | first postoperative night
  The primary objective is to compare postoperative sleep quality, as measured using a bispectral index-Vista monitor during the first night after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes